CLINICAL TRIAL: NCT02554344
Title: Effect of Curcumin in Treatment of Squamous Cervical Intraepithelial Neoplasias (CINs)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: no subject accrual
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 015-074
Record Dates: First submitted 2015-09-14; First posted 2015-09-18 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: CIN3; Squamous CIN3
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Patients (Experimental): Fourteen subjects with histologically confirmed squamous CIN3 will be enrolled in a single arm study. All patients will receive 500 mg of curcumin administered orally, twice a day for 12 weeks upon enrollment on trial.
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin — Patients will receive 500mg of curcumin administered orally, twice a day for 12 weeks.
  Other Names: Turmeric; BCM-95®

SUMMARY:
The purpose of this study is to determine the safety, feasibility, and regression rate of using curcumin in patients with Cervical Intraepithelial neoplasias (CIN3). The secondary objectives of this study is to evaluate patients with CIN3 for the presence of high-risk Human papillomavirus (HPV) and to perform an inflammatory panel on dysplasia biopsies from patients with CIN3 to determine which factors play a role in persistence of CIN3.

DETAILED DESCRIPTION:
Fourteen women with a biopsy-confirmed CIN3 diagnosis will be enrolled. The participants will receive 500mg of curcumin orally twice daily for 12 weeks. Colposcopies will be performed at the participants' baseline, 6 week, and 12 week visits. Two biopsies will be performed at the baseline and 12 week visit, and if there is suspicion for cancer formation or invasion, at the 6-week visit. One sample will be used for histologic examination, while the other sample will be used for p65 assays. Based on the biopsy, if cancer is present, then the patient will be referred to gynecologic oncology for further care and the trial will be terminated. At the end of the 12 week period, if CIN3 persists, Loop electrosurgical excision procedure (LEEP) or Cold knife conisation (CKC) will be performed to remove the dysplastic cells as this is considered standard of care.

ELIGIBILITY:
Inclusion Criteria: A patient will be eligible for inclusion in this study if she meets all of the following criteria:

1. The patient must be 21 or older and able to give informed consent.
2. Patient must have histologically confirmed squamous CIN3.
3. There must be an adequate colposcopy.
4. Patient must have no abnormal cells in their endocervical curettage (ECC).
5. There must be no suspicion of invasion.

Exclusion Criteria: A patient will be ineligible for inclusion in this study if she meets any of the following criteria:

1. Women who are pregnant or lactating.
2. HIV+ status
3. Adenocarcinoma in situ or any invasive cancer of the cervix.
4. Gallstones or bile duct obstructions.
5. Patients on anti-coagulant/anti-platelet therapies.
6. Patients on immunosuppressive therapies.
7. Patients may not receive any other investigational treatments while participating in this study.
8. Concurrent severe, uncontrolled infection or intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Determine the safety and feasibility using curcumin in patients with CIN3 where toxicities will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. | 4 months
  Events will be recorded from the time of informed consent signature through the 30 days following the last study treatment.

SECONDARY OUTCOMES:
Regression Rate | 4 months
  Determine if treatment with oral curcumin for 12 weeks will cause regression of CIN3. The response will be measured based on histology of the tissue. The location of CIN3 will be documented in the case report form. The degree of CIN3 will be recorded visually as well as histologically through biopsy. The total area will be estimated by the physicians and tissue sections will be made and the degree of dysplasia will be determined.
Overall Response | 4 months
  Recorded from the start of the treatment until disease progression/recurrence. The patient's best response assignment will depend on the finding of target disease and will also take into consideration the appearance of new lesions.
Pathologic Response | 4 months
  Patients will undergo colposcopy followed by LEEP or CKC if residual dysplasia is still present after treatment. Using standard morphologic criteria, the biopsies will be evaluated, dysplasia will be graded.
Rate of patients in which p65, phosphorylated p65, and acetylated p65 play a role in the persistence of CIN. | 4 months
  The minced tissue will be homogenized using a Dounce homogenizer and and centrifuged at 16,000 × g at 4 °C for 10 min. The proteins will be fractionated by SDS-PAGE, electrotransferred to polyvinylidene fluoride (PVDF) membranes, blotted with each antibody sequentially (p65, phosphorylated p65, or acetylated p65; Cell Signaling Technology; Danvers, MA), and detected by enhanced chemiluminescence (Amersham ECL Advance kit; GE Healthcare Life Sciences, Inc, Piscataway, NJ). The PVDF filters will be stripped and re-probed so each blot can be used to measure all three antibodies on the same samples.
Evaluation of patients with CIN3 for the presence of high-risk HPV. | 4 months
  HPV tests will be conducted using the AMPLICOR® Human Papillomavirus Test. This is a polymerase chain reaction-based (PCR) qualitative test for the detection of 13 high-risk HPV geneotypes most commonly associated with cervical pre-cancer, including HPV-16 and -18.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Matthews, MD, Principal Investigator — Baylor Research Institute/Texas Oncology
Locations (1):
- Baylor Charles A. Sammons Cancer Center, Dallas, Texas, United States